CLINICAL TRIAL: NCT01371071
Title: Clinically Isolated Syndrome and Newly Diagnosed Multiple Sclerosis: Diagnostic, Prognostic and Therapy - Response Markers - a Prospective Observational Study (Berlin CIS-COHORT)
Brief Title: Cohort Study of Clinically Isolated Syndrome and Early Multiple Sclerosis
Acronym: CIS-COHORT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Friedemann Paul, MD; Klemens Ruprecht, MD; Judith Bellmann-Strobl, MD, Charité - Universiätsmedizin Berlin
Other Study IDs: EK1/2011
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Sclerosis, MS; Clinically Isolated Syndrome
Keywords: Clinically isolated syndrome (CIS); Multiple sclerosis (MS); Immunomodulatory therapy; Prognostic markers; MRI; OCT
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples (serum and plasma, with DNA), urine, saliva, CSF (if routine lumbar puncture was performed, no additional lumbar punctures for the study)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CIS or early relapsing-remitting MS

SUMMARY:
A majority of patients with multiple sclerosis initially presents with a single demyelinating event, e.g. in the optic nerves, brain, brainstem or spinal cord, referred to as a clinically isolated syndrome (CIS). Not all patients with CIS get a relapse and develop multiple sclerosis but in those patients who do, irreversible damage of the central nervous system, e.g. axonal damage, is already detectable in that early stage of disease. Early initiation of immunomodulatory therapy is crucial for patients with clinically isolated syndrome who are at high risk for the development of multiple sclerosis. Vice versa identification of low risk patients could help to avoid an unnecessary therapy. In this prospective observational study we want to follow up patients with CIS and early multiple sclerosis over a period of four years and obtain clinical, laboratory and MRI - data in order to identify risk factors for relapses, prognostic factors and therapy response markers.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* signed informed consent
* clinically isolated syndrome within the last 6 months
* diagnosis of multiple sclerosis within the last two years

Exclusion Criteria:

* eye disease that could interfere with OCT (e.g. glaucoma, diabetic retinopathy)
* secondary progressive multiple sclerosis
* pregnancy
* contraindications for MRI, e.g. pacemaker, metal implants, allergy against gadolinium
* alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruted at neurological outpatient clinics and neurologcial clinics of the charité and neurologists' medical practices.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
time (in days) until relapse during the observation period of four years | 48 months

SECONDARY OUTCOMES:
MRI - parameters: number and volume of T2 and gadolinium enhancing lesions, analysis of lesion patterns (spinal und cerebral MRI) | 48 months
biomarkers: RNA, microRNA, DNA, proteins, enzymes, autoantibodies, antiviral antibodies, virus DNA, Vitamin D and lipids in serum, plasma, peripheral cells, urine, saliva and CSF | 48 months
Optical Coherence Tomography (OCT): thickness of the retinal nerve fibre layer (RNFL) or total macular volume (TMV) | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Prof., Principal Investigator — Charite - Universitätsmedizin Berlin; Klemens Ruprecht, Dr., Principal Investigator — Charite University, Berlin, Germany; Judith Bellmann-Strobl, Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Department of Neurology, Charité - Universitätsmedizin Berlin, Berlin
  - NeuroCure Clinical Research Center, Charité - Universitätsmedizin Berlin, Berlin

REFERENCES:
- [Derived] Gottwald NS, Asseyer S, Chien C, Brasanac J, Nauman AT, Rust R, Schmitz-Hubsch T, Strobl JB, Ruprecht K, Paul F, Regitz-Zagrosek V, Gold SM, Sperber PS. Impact of sex on clinical outcome in early Multiple Sclerosis. Mult Scler Relat Disord. 2024 Aug;88:105749. doi: 10.1016/j.msard.2024.105749. Epub 2024 Jun 29. PMID 38959589
- See also: Homepage of the NeuroCure Clinical Research Center — http://www.neurocure.de